CLINICAL TRIAL: NCT00001341
Title: A Phase I Trial of ZD1694 (TOMUDEX® (Registered Trademark)), an Inhibitor of Thymidylate Synthase, in Pediatric Patients With Advanced Neoplastic Disease
Brief Title: A Phase I Trial of ZD1694 (TOMUDEX), an Inhibitor of Thymidylate Synthase, in Pediatric Patients With Advanced Neoplastic Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 930210; 93-C-0210
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-08

CONDITIONS: Neoplasm
Keywords: Antifolate; Inhibitor; Pharmacokinetics; Thymidylate Synthetase; Toxicity
MeSH Terms: conditions — Neoplasms | interventions — raltitrexed

INTERVENTIONS:
Drug: ZD1694 (TOMUDEX)

SUMMARY:
Thymidylate synthase (TS), an enzyme which acts by utilizing 5,10-CH(2)FH(4) in the reductive methylation of deoxyuridylate (dUMP), is required for the de novo synthesis of thymidylate and is a potential chemotherapeutic target. ZD1694 is a new quinazolone folate analog that directly inhibits TS. This phase I trial and pharmacokinetic study will describe and define the toxicities, determine the MTD, and describe the plasma pharmacokinetics of ZD1694 in pediatric patients with refractory cancer. The starting dose for this trial will be 2.0 mg/m(2) administered as a 15 minute IV infusion every 21 days.

DETAILED DESCRIPTION:
Thymidylate synthase (TS), an enzyme which acts by utilizing 5,10-CH(2)FH(4) in the reductive methylation of deoxyuridylate (dUMP), is required for the de novo synthesis of thymidylate and is a potential chemotherapeutic target. ZD1694 is a new quinazolone folate analog that directly inhibits TS. This phase I trial and pharmacokinetic study will describe and define the toxicities, determine the MTD, and describe the plasma pharmacokinetics of ZD1694 in pediatric patients with refractory cancer. The starting dose for this trial will be 2.0 mg/m(2) administered as a 15 minute IV infusion every 21 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Histologically proven malignancy considered refractory to standard therapy. Objective evidence of progression on prior therapy required.

No leukemia.

Bone marrow involvement by tumor acceptable. Marrow biopsy required if there is a history of involvement or peripheral counts are inadequate.

PRIOR/CONCURRENT THERAPY:

Biologic Therapy: Recovery from toxic effects of prior immunotherapy required.

Chemotherapy: No more than 2 prior chemotherapy regimens and recovered. At least 2 weeks since myelosuppressive therapy (6 weeks since nitrosoureas).

Endocrine Therapy: Not specified.

Radiotherapy:

No prior central axis irradiation (i.e., skull, spine, ribs, pelvis).

Recovery from toxic effects of prior radiotherapy required.

Surgery: Not specified.

Other: No prior bone marrow transplantation.

PATIENT CHARACTERISTICS:

Age: 21 and under.

Performance status: ECOG 0-2.

Life expectancy: At least 8 weeks.

Hematopoietic:

(unless histologic evidence of bone marrow involvement by tumor).

AGC at least 1,500/mm3.

Platelet count at least 100,000/mm3.

Hemoglobin at least 8.0 g/dL.

Prior transfusion acceptable.

Hepatic:

Bilirubin no greater than 2 times normal.

ALT no greater than 2 times normal.

Renal:

Creatinine less than 1.5 mg/dL OR

Creatinine clearance greater than 60 mL/min/1.73 sqm.

Cardiovascular: Not specified.

Pulmonary: Not specified.

OTHER:

No significant accumulation of third space fluid.

No significant systemic illness (e.g., infection).

No pregnant or nursing women.

Pregnancy test required in fertile women.

All patients or their guardians must sign an informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1993-09; Study Completion 2001-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Jackman AL, Taylor GA, Gibson W, Kimbell R, Brown M, Calvert AH, Judson IR, Hughes LR. ICI D1694, a quinazoline antifolate thymidylate synthase inhibitor that is a potent inhibitor of L1210 tumor cell growth in vitro and in vivo: a new agent for clinical study. Cancer Res. 1991 Oct 15;51(20):5579-86. PMID 1913676
- [Background] Jackman AL, Marsham PR, Moran RG, Kimbell R, O'Connor BM, Hughes LR, Calvert AH. Thymidylate synthase inhibitors: the in vitro activity of a series of heterocyclic benzoyl ring modified 2-desamino-2-methyl-N10-substituted-5,8-dideazafolates. Adv Enzyme Regul. 1991;31:13-27. doi: 10.1016/0065-2571(91)90006-8. PMID 1877386
- [Background] Cunningham D, Zalcberg JR, Rath U, Olver I, Van Cutsem E, Svensson C, Seitz JF, Harper P, Kerr D, Perez-Manga G, et al. 'Tomudex' (ZD1694): results of a randomised trial in advanced colorectal cancer demonstrate efficacy and reduced mucositis and leucopenia. The 'Tomudex' Colorectal Cancer Study Group. Eur J Cancer. 1995 Nov;31A(12):1945-54. doi: 10.1016/0959-8049(95)00502-1. PMID 8562146